CLINICAL TRIAL: NCT04819360
Title: Injections of Botulinum Toxin a or Anticholinergic Treatment As First Line Therapy to Treat Neurogenic Overactive Bladder in Patients with Multiple Sclerosis
Brief Title: Botulinum Toxin a Vs Anticholinergic Treatment of Neurogenic Overactive Bladder in Patients with Multiple Sclerosis
Acronym: SEPTOX
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Brigitte Schürch (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Sponsor-Investigator, Brigitte Schürch, Professor, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEPTOX
Record Dates: First submitted 2020-12-13; First posted 2021-03-26 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2022-02

CONDITIONS: Urinary Bladder, Neurogenic; Multiple Sclerosis
Keywords: Botulinum toxin; Neurogenic bladder; Multiple sclerosis; Anticholinergic drugs
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Multiple Sclerosis | interventions — Solifenacin Succinate; Tablets; Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vesicare (Active Comparator): Group 1: will be treated with an anticholinergic (Vesicare® 10 mg per day for 12 weeks)
  Interventions: Drug: VESIcare 10Mg Tablet
- Botox (Active Comparator): Group 2: will receive an intra-detrusor injection of a low dose of botulinum toxin type A (100 U of BOTOX®).
  Interventions: Drug: Botox 100 UNT Injection

INTERVENTIONS:
Drug: VESIcare 10Mg Tablet — Vesicare® 10 mg per day for 12 weeks
  Vesicare 10mg 12 weeks
  Other Names: Vesicare
  Arms: Vesicare
Drug: Botox 100 UNT Injection — 1 injection of Botox® 100 UNT
  Other Names: Botox
  Arms: Botox

SUMMARY:
Botulinum toxin type A injections into the detrusor at a dose of 200 units (U) of BOTOX® are a recognized second-line treatment for the treatment of adult neurogenic lower urinary tract disorders. Anticholinergics are established as the usual first-line treatment for neurogenic detrusor hyperactivity, but are oft not sufficiently effective and have significant side effects. In patients with multiple sclerosis (MS) suffering from overactive bladder, the 200 U dose of BOTOX® is very effective but induces a risk of urinary retention in 30% of patients requiring the temporary use of self-catheterization1. At 100 U, a recent study shows the efficacy and very good tolerance of botulinum toxin A in terms of probing risk in MS patients with overactive bladder and failure of anticholinergics. Furthermore, the efficacy of anticholinergics in MS has been little studied and is also disputed.

The investigators plan to test the therapeutic alternative as the first line of treatment in two groups of randomized MS patients from a homogeneous population suffering from overactive bladder:

* a group testing the effectiveness of low doses of botulinum toxin type A (100 U, BOTOX®),
* the other group receiving the standard anticholinergic treatment (solifenacin succinate, Vesicare®).

During this pilot study, the efficacy and side effects profile of each treatment will be analyzed in order to determine the amplitudes of effect and the safety profiles in this population and in order to establish the statistical hypotheses for a subsequent randomized multicenter study. The aim of this study will be to establish the benefit of botulinum toxin at a dose of 100 U as a first-line treatment instead of anticholinergics

DETAILED DESCRIPTION:
Botulinum toxin type A (BOTOX®) injections will performed on an outpatient basis by cystoscopy under local anesthesia. Twenty minutes after an intravesical instillation of 20 ml of 0.2% ropivacaine, the botulinum toxin is injected into the detrusor muscle using a flexible injection needle at a rate of 10 U of BOTOX® per mL (10 points of 1 mL injections). Intravenous prophylaxis (cefuroxime 1.5 g) will be performed 30 minutes before the injections.

Patients in the Vesicare® arm will be given the tablets at the baseline visit to be taken once a day in the morning for 12 weeks. For this arm, there will be no antibiotic prophylaxis.

Randomization will be carried out via eCRF in the secuTrial® environment with an integrated Interactive Web Response System (IWRS) function allowing the allocation of a participant to one of the two intervention groups. Randomization will be carried out using a randomization table in blocks of 2, predefined without the knowledge of the investigator, respecting a balanced allocation between the two groups, necessary given the modest number of participants in the study.

The intensity of therapeutic responses for each treatment is not precisely known in this patient population. As a result, there are no reliable preliminary data which would allow the investigators to calculate under these "effect size" assumptions the necessary numbers of participants to be randomized between the two intervention groups in order to demonstrate a possible superiority of treatment by injection of BOTOX® 100 U in comparison to the reference anticholinergic treatment. The comparative study will therefore only be accessible after determining the intensity of these effects.

Within the framework of a pilot study not directly comparative of the therapeutic approaches but seeking to identify the amplitude of the effects obtained independently by the two treatments, it does not appear necessary to resort to a study design with "double-dummy" to leave the patient blind to the method used. Such an approach would require the use of a sham injection by cystoscopic route in the group treated with anticholinergics and would not appear ethical in this context.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple sclerosis (MS) with neurogenic detrusor overactivity proven by urodynamics
* Stable MS with an Expanded Disability Severity Score (EDSS) less than or equal to 6.5
* Voluntary micturitions
* Number of micturitions > 8 per day, with or without episodes of urgency and urgency incontinence
* Signed informed consent form

Exclusion Criteria:

* Pregnancy, breastfeeding
* Patients requiring self-catheterizations
* Patients unable or unwilling to learn self-catheterisation
* Recent (<12 weeks) or current treatment with botulinum toxin for any non-urological indication
* Recent (≤ 8 weeks) or current treatment with anticholinergic drugs
* Patients with a positive history or evidence of pelvic / urological abnormality (interstitial cystitis, bladder lithiasis in the 6 months preceding the screening, or any other condition / operation affecting the bladder or prostate)
* Any contraindication to Vesicare®:

  * Hypersensitivity to the active ingredient or to one of the excipients
  * Urinary retention
  * Untreated narrow-angle glaucoma
  * Severe gastrointestinal illness (e.g. toxic megacolon)
  * Myasthenia gravis
  * Severe hepatic failure
  * Hemodialysis
  * Severe renal failure, or liver function disturbances of moderate severity with concomitant treatment with a strong inhibitor of the CYP3A4 isoenzyme, including patients at risk for these diseases.
* Any contraindication to BOTOX®:

  * Known hypersensitivity to the active substance or to one of the excipients
  * Presence of a symptomatic infection at the planned injection site(s)
  * Urinary tract infection at the time of planned treatment
  * Patients who present with acute urinary retention at the time of treatment and who do not regularly use bladder catheterization
  * Patients who do not want and / or cannot, if necessary, perform self-intermittent catheterisation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2024-04-21 (Actual)

PRIMARY OUTCOMES:
Magnitude of effect - Number of micturitions per 24h | 6 weeks
  The difference in mean values of [the number of micturitions / 24 h for the last 3 days] at T0 (inclusion) and T6W (6 weeks after start of the treatment).

SECONDARY OUTCOMES:
Other parameters of effects - Number of urgent urinations per 24h | 2, 6 and 12 weeks after treatment start
  The difference in mean values of [the number of episodes of urgent urination / 24 h for the last 3 days] at T0 (inclusion) and T2W (2 weeks after start of the treatment).
  The difference in mean values of [the number of episodes of urgent urination / 24 h for the last 3 days] at T0 (inclusion) and T6W (6 weeks after start of the treatment).
  The difference in mean values of [the number of episodes of urgent urination / 24 h for the last 3 days] at T0 (inclusion) and T12W (12 weeks after start of the treatment).
Other parameters of effects - Number of urgency urinary incontinence episodes per 24h | 2, 6 and 12 weeks after treatment start
  The difference in mean values of [the number of urgency urinary incontinence episodes / 24 h for the last 3 days] at T0 (inclusion) and T2W (2 weeks after start of the treatment).
  The difference in mean values of [the number of urgency urinary incontinence episodes / 24 h for the last 3 days] at T0 (inclusion) and T6W (6 weeks after start of the treatment).
  The difference in mean values of [the number of urgency urinary incontinence episodes / 24 h for the last 3 days] at T0 (inclusion) and T12W (12 weeks after start of the treatment).
Other parameters of effects - Number of nocturnal micturition episodes per 24h | 2, 6 and 12 weeks after treatment start
  The difference in mean values of [the number of nocturnal micturition episodes / 24 h for the last 3 days] at T0 (inclusion) and T2W (2 weeks after start of the treatment).
  The difference in mean values of [the number of nocturnal micturition episodes / 24 h for the last 3 days] at T0 (inclusion) and T6W (6 weeks after start of the treatment).
  The difference in mean values of [the number of nocturnal micturition episodes / 24 h for the last 3 days] at T0 (inclusion) and T12W (12 weeks after start of the treatment).
Other parameters of effects - Number of 100% dry patients | 6 and 12 weeks after treatment start
  The difference in mean values of [the number of 100% dry patients / 24 h for the last 3 days] at T0 (inclusion) and T6W (6 weeks after start of the treatment).
  The difference in mean values of [the number of 100% dry patients / 24 h for the last 3 days] at T0 (inclusion) and T12W (12 weeks after start of the treatment).
Other parameters of effects - Urodynamic parameter : cystomanometric capacity | 6 weeks after treatment start
  The difference in cystomanometric capacity at 6 weeks after the start of the treatment, as compared to inclusion values.
Other parameters of effects - Urodynamic parameter : reflex volume at first contraction | 6 weeks after treatment start
  The difference in reflex volume at first contraction at 6 weeks after the start of the treatment, as compared to inclusion values.
Other parameters of effects - Urodynamic parameter : bladder compliance | 6 weeks after treatment start
  Bladder compliance describes the relationship between change in bladder volume (ΔV) and change in detrusor pressure (Δpdet).
  Compliance is calculated by dividing the volume change (∆V) by the change in detrusor pressure (∆pdet) during that change in bladder volume (C= ΔV/∆pdet). It is expressed in ml/cm H2O.
Other parameters of effects - Urodynamic parameter : maximum detrusor pressure | 6 weeks after treatment start
  The difference in maximum detrusor pressure at 6 weeks after the start of the treatment, as compared to inclusion values.
Other parameters of effects - Urodynamic parameter : post-void residual after flowmetry | 6 weeks after treatment start
  The difference in post-void residual after flowmetry at 6 weeks after the start of the treatment, as compared to inclusion values.

OTHER OUTCOMES:
Patients reported outcomes - Patients' satisfaction | 2, 6 and 12 weeks
  Patients' satisfaction, measured by the Patient Global Impression of Improvement (PGI-I), at 2, 6 and 12 weeks after the start of the treatment, as compared to inclusion values.
Patients reported outcomes - Patients' specific quality of life | 2, 6 and 12 weeks
  Patients' specific quality of life, measured by the Urinary Incontinence Quality of Life Scale (I-QOL), at 2, 6 and 12 weeks after the start of the treatment, as compared to inclusion values.
Patients reported outcomes - Subjective improvement | 2, 6 and 12 weeks
  Patients' subjective improvement, measured by a Visual Analog Scale (VAS), at 2, 6 and 12 weeks after the start of the treatment, as compared to inclusion values.
Security - Self-catheterizations | Any time during the 12 weeks of the trial
  Need for self-catheterizations according to pre-specified criteria, at any time during the trial
Security - Urinary tract infections | Any time during the 12 weeks of the trial
  Number of urinary tract infections episodes, at any time during the trial
Security - Adverse drug reactions due to anticholinergic drugs | Any time during the 12 weeks of the trial
  Number of adverse drug reactions due to anticholinergic drugs, at any time during the trial
Security - Adverse drug reactions due to Botox | Any time during the 12 weeks of the trial
  Number of adverse drug reactions due to Botox, at any time during the trial

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Schürch, Prof., Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chermansky C, Schurch B, Rahnama'i MS, Averbeck MA, Malde S, Mancini V, Valentini F, Sahai A. How can we better manage drug-resistant OAB/DO? ICI-RS 2018. Neurourol Urodyn. 2019 Dec;38 Suppl 5:S46-S55. doi: 10.1002/nau.24055. PMID 31821628